CLINICAL TRIAL: NCT04830306
Title: Comparison of Submaximal Exercise Tests With Maximal Exercise Test
Brief Title: Step, Walk, Bike: Comparisons of Fitness Assessments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00108027
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2021-11

CONDITIONS: Cardiorespiratory Fitness
Keywords: aerobic power; CPET; CPEX; cardiopulmonary exercise testing; exercise capacity; functional capacity; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All subjects will be asked to complete the three exercise tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 6MST (Active Comparator): Six minute step test
  Interventions: Behavioral: Exercise
- 6MWT (Active Comparator): Six minute walk test
  Interventions: Behavioral: Exercise
- CPET (Active Comparator): Cardiopulmonary exercise test
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Completion of exercise in accordance with assigned protocol

SUMMARY:
To compare cardiorespiratory fitness parameters (oxygen consumption and respiratory ventilation) measured during two sub-maximal exercise tests (six minute step test, 6MST & six minute walk test, 6 MWT) with maximal exercise test (cardiopulmonary exercise test, CPET)

DETAILED DESCRIPTION:
After enrollment, the subjects will complete each of the following CRF assessments:

Sub-maximal exercise test Six Minute Step Test (6MST): A face mask with the VO2 Master expired gas analysis device will be secured in position with head strap. Subjects will rest seated for 5 minutes prior to the start of the test. The subject will be given a standardized set of instructions on how to complete the test by raising each knee to 90 degrees of hip flexion. The total number of steps completed during the timed 6-minute period will be recorded.

Sub-maximal exercise test Six Minute Walk Test (6MWT): A face mask with the VO2 Master expired gas analysis device will be secured in position with head strap. Subjects will rest seated for 5 minutes prior to the start of the test. A 30-m unobstructed hallway with turning points marked with small cones will be used. The subject will be given a standardized set of instructions on how to complete the test. The total distance walked during the timed 6-minute period will be recorded.

Maximal exercise cardiopulmonary exercise test (CPET): The CPET is performed using an electromagnetically-braked cycle ergometer, 12-lead continuous ECG, continuous pulse oximetry, continuous expired gas analysis (oxygen and carbon dioxide) with ventilation [termed 'metabolic cart'] and intermittent non-invasive blood pressure measurement every 2 minutes. Once the subject is seated comfortably on the bike and adjusted for optimum cycling position, the face mask is fitted. The subjects are instructed on how to perform the incremental ramp test, starting with a baseline rest phase (no leg turnover) for 2 mins followed by reference phase of 2 mins of leg turnover with no resistance (0 watts). The incremental rise in work-rate from baseline is pre-determined by using the equation derived by Wasserman and colleagues in which the same work-rate is increased throughout the test to the limit of tolerance. A work-rate is selected by study staff to aim for a test duration of between 8 and 12 minutes. The subjects are instructed to maintain a cycling cadence of 55 - 65 revolutions per minute (rpm) during the exercise phase. One the limit of tolerance (maximal watts) is reached the resistance on the bike is removed () watts) and the subjects are encouraged to continue cycling for a further 2 mins during the recovery phase.

The order in which 6MST and 6MWT are performed will be randomized. Between test the subjects will be allowed to rest in a chair until the heart rate is within 5 beats per min of resting values and blood pressure in within 10 mmHg of resting values. The CPET will be conducted once both 6MWT and 6MST have been completed. If the subject expresses fatigue after either 6MWT and 6MST, then the subject may elect to re-attend on a separate day to complete the evaluation. At completion of exercise evaluations the subjects will be discharged from study participation. No further follow up will be performed.

Up to 40 subjects aged 18 or older will be enrolled.

Inclusion Criteria:

* Age 18 and older
* Able to speak English
* Ambulatory [assistive devices ok]
* Able to provide informed consent

Exclusion Criteria:

* Any exclusion criteria listed in table 8 American Thoracic Society /American College of Chest Physicians Statement on CPET
* Inmate of correctional facility (i.e. prisoner)
* Diagnosed history of dementia
* Inability to ambulate independently
* Considered inappropriate to participate by Principal Investigator

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Able to speak English
* Ambulatory [assistive devices ok]
* Able to provide informed consent

Exclusion Criteria:

* Any exclusion criteria listed in table 8 American Thoracic Society /American College of Chest Physicians Statement on CPET
* Inmate of correctional facility (i.e. prisoner)
* Diagnosed history of dementia
* Inability to ambulate independently
* Considered inappropriate to participate by Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Total amount of oxygen consumed per minute as measured by wearable face mask | Up to 15 minutes
  Oxygen measured in mL/min

SECONDARY OUTCOMES:
Total amount of respiratory ventilation per minute as measured by wearable face mask | Up to 15 minutes
  Respiratory ventilation measured in liters per minute

CONTACTS AND LOCATIONS:
Overall Officials: David MacLeod, FRCA, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No